CLINICAL TRIAL: NCT07396246
Title: The HIPE RCT - Comparison Between Transarterial Musculoskeletal Embolization (TAME) and Platelet-Rich Plasma (PRP) Injection for the Treatment of Greater Trochanteric Pain Syndrome - A Randomized Controlled Trial
Brief Title: Comparison Between Transarterial Musculoskeletal Embolization and Platelet-Rich Plasma Injection for the Treatment of Greater Trochanteric Pain Syndrome
Acronym: HIPE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Unidade Local de Saúde do Alto Ave, EPE (Other)
Collaborators: Serviço de Ortopedia da ULS Alto Ave (Unknown); Serviço de Imagiologia da ULS Alto Ave (Unknown)
Responsible Party: Principal Investigator, Pedro Lopes, Interventional Radiologist, Unidade Local de Saúde do Alto Ave, EPE
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114-2025 CAF
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-09

CONDITIONS: Trochanteric Syndrome
Keywords: Embolization; Musculoskeletal; Hip; Greater Trochanter Pain Syndrome; Pain management; PRP
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transarterial Musculoskeletal Embolization (Active Comparator): Participants assigned to this arm will undergo transarterial musculoskeletal embolization (TAME) under local anesthesia. The procedure will be performed by an experienced interventional radiologist using selective catheterization of pathological peri-trochanteric vessels supplying the affected hip structures. Embolization will be carried out using a temporary, reabsorbable embolic microsphere (Nexsphere-F®, CE approved) to achieve transient vessel occlusion. The aim of the procedure is to reduce pathological neovascularization and inflammation associated with Greater Trochanteric Pain Syndrome.
  Interventions: Procedure: Transarterial Musculoskeletal Embolization
- Platelet-Rich Plasma Injection (Active Comparator): Participants assigned to this arm will receive a single ultrasound-guided intratendinous injection of autologous platelet-rich plasma (PRP) into the affected gluteal tendon. The procedure will be performed by an orthopedic hip specialist under sterile conditions. PRP will be prepared from the participant's own blood using a standardized centrifugation protocol. The objective of this intervention is to promote tendon healing and reduce pain and functional impairment associated with Greater Trochanteric Pain Syndrome.
  Interventions: Biological: Platelet-Rich Plasma Injection

INTERVENTIONS:
Procedure: Transarterial Musculoskeletal Embolization — Transarterial musculoskeletal embolization (TAME) is performed under local anesthesia by an experienced interventional radiologist. The procedure consists of selective catheterization and embolization of pathological peri-trochanteric vessels supplying the affected hip structures. A temporary, reabsorbable embolic microsphere (Nexsphere-F®, CE approved) is used to achieve transient vessel occlusion, with the objective of reducing pathological neovascularization and inflammation associated with Greater Trochanteric Pain Syndrome.
  Other Names: TAME
  Arms: Transarterial Musculoskeletal Embolization
Biological: Platelet-Rich Plasma Injection — Platelet-rich plasma (PRP) injection consists of a single ultrasound-guided intratendinous administration of autologous PRP into the affected gluteal tendon. PRP is prepared from the participant's own blood using a standardized centrifugation protocol and injected under sterile conditions by an orthopedic hip specialist. The intervention aims to promote tendon healing and reduce pain and functional impairment associated with Greater Trochanteric Pain Syndrome.
  Other Names: PRP injection
  Arms: Platelet-Rich Plasma Injection

SUMMARY:
Greater Trochanteric Pain Syndrome (GTPS) is a common cause of lateral hip pain that can significantly affect daily activities and quality of life. Standard treatments include physical therapy, anti-inflammatory medications, and local injections, but many patients continue to experience persistent symptoms.

This randomized controlled trial aims to compare two minimally invasive treatment options for GTPS: transarterial musculoskeletal embolization (TAME) and platelet-rich plasma (PRP) injection. Participants will be randomly assigned to receive either TAME or PRP.

The main goal of the study is to evaluate which treatment is more effective in reducing pain. Secondary goals include comparing functional improvement, quality of life, and safety between the two treatments. Pain and functional outcomes will be assessed at baseline and during follow-up at 1, 3, 6, and 12 months after treatment.

This study seeks to provide evidence on the effectiveness and safety of TAME compared with PRP injection for patients with Greater Trochanteric Pain Syndrome.

DETAILED DESCRIPTION:
This is a prospective, single-center, parallel-group randomized controlled trial designed to compare the efficacy and safety of transarterial musculoskeletal embolization (TAME) versus platelet-rich plasma (PRP) injection in patients with Greater Trochanteric Pain Syndrome (GTPS).

Eligible adult patients with clinically and radiologically confirmed GTPS and persistent symptoms despite at least three months of conservative treatment will be enrolled. Participants will be randomized in a 1:1 ratio to receive either TAME or PRP injection.

TAME will be performed under local anesthesia by an experienced interventional radiologist, using selective catheterization and embolization of pathological vessels supplying the affected peri-trochanteric structures. A temporary, reabsorbable embolic agent (Nexsphere-F®, CE approved) will be used to achieve a transient embolization effect aimed at reducing pathological neovascularization and inflammation.

PRP treatment will consist of a single ultrasound-guided intratendinous injection of autologous platelet-rich plasma into the affected gluteal tendon, performed by an orthopedic hip specialist under sterile conditions.

This is a single-blind study. A trained nurse from the radiology department, blinded to treatment allocation, will conduct all follow-up assessments and collect outcome data to minimize assessment bias.

The primary outcome measure is pain reduction assessed using the Visual Analog Scale (VAS) at baseline and at 1, 3, 6, and 12 months after treatment. Secondary outcome measures include functional improvement assessed using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), quality of life evaluated with the EQ-5D-5L questionnaire, and the incidence of adverse events graded according to the CIRSE adverse event classification system.

A total of 30 participants (15 per group) will be included. Patients who do not achieve at least a 50% reduction in pain at 12 months will be eligible to cross over to the alternative treatment arm.

Statistical analysis will include descriptive statistics for baseline characteristics and outcomes. Group comparisons will be performed using independent t-tests or chi-square tests as appropriate. Longitudinal changes will be analyzed using repeated measures analysis of variance or mixed-effects models. Statistical significance will be set at p < 0.05.

The study will be conducted in accordance with the Declaration of Helsinki and Good Clinical Practice guidelines. Ethics approval has been obtained from the Unidade Local de Saúde do Alto Ave ethics committee. Written informed consent will be obtained from all participants prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GTPS confirmed by clinical and imaging assessments
* Persistent symptoms despite at least 3 months of conservative treatment (e.g., physical therapy, NSAIDs)
* Willingness to participate and provide informed consent
* Availability for follow-up assessments at 1, 3, 6, and 12 months post-treatment

Exclusion Criteria:

* Prior hip surgery or other interventions (e.g., joint replacement, prior PRP injections or embolization)
* Severe osteoarthritis (Tonnis III)
* Active lumbar radiculopathy with pain, numbness, or weakness in a dermatomal distribution
* Contraindications for PRP injections (e.g., active infection, coagulopathy, antiplatelet or anticoagulation therapy,
* Pregnancy or breastfeeding
* Severe comorbidities that would interfere with participation
* Active cancer or other malignancies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain reduction assessed by Visual Analog Scale (VAS) | Baseline, 1 month, 3 months, 6 months, and 12 months after treatment
  Change in pain intensity from baseline measured using the Visual Analog Scale (VAS), comparing participants treated with transarterial musculoskeletal embolization (TAME) versus platelet-rich plasma (PRP) injection.

SECONDARY OUTCOMES:
Functional improvement assessed by WOMAC score | Baseline, 1 month, 3 months, 6 months, and 12 months after treatment
  Change in functional status from baseline measured using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), comparing participants treated with transarterial musculoskeletal embolization (TAME) versus platelet-rich plasma (PRP) injection.
Quality of life assessed by EQ-5D-5L questionnaire | Baseline, 1 month, 3 months, 6 months, and 12 months after treatment
  Change in health-related quality of life from baseline measured using the EQ-5D-5L questionnaire, comparing participants treated with transarterial musculoskeletal embolization (TAME) versus platelet-rich plasma (PRP) injection.
Incidence of adverse events related to TAME or PRP | From treatment to 12 months after the procedure
  Number and severity of procedure-related adverse events associated with transarterial musculoskeletal embolization (TAME) or platelet-rich plasma (PRP) injection, graded according to the CIRSE adverse event classification system.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro M M Lopes, MD, Principal Investigator — Unidade Local de Saúde do Alto Ave
Locations (1):
- Unidade Local de Saúde do Alto Ave, Guimarães, Portugal

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results of this study, including baseline characteristics and outcome measures (VAS, WOMAC, EQ-5D-5L, and adverse events), will be made available for secondary research purposes.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From 6 months after publication of the primary results to 5 years thereafter.
Access Criteria: Access to de-identified individual participant data and supporting documents will be granted to qualified researchers upon reasonable request. Requests must include a research proposal and statistical analysis plan and will be reviewed by the study investigators. Data will be shared for non-commercial scientific research purposes only and under a data use agreement.